CLINICAL TRIAL: NCT03474861
Title: A Combination Study to Evaluate the Safety and Efficacy of an Anticancer Medication (A01) With Immune Cells (IC01) in Subjects With Advanced Gastrointestinal Cancer
Brief Title: Safety and Efficacy of an Anticancer Medication Combined With Immune Cells in Subjects With Gastrointestinal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangzhou Converd Co., Ltd. (Industry)
Collaborators: The Second Hospital of Jia Xing (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVD20180401002
Record Dates: First submitted 2018-03-07; First posted 2018-03-23 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy (Experimental): The subjects will be given combination therapy which consists of an anticancer medication (A01) and immune cells (IC01).
  Interventions: Biological: anticancer medication A01; immune cells IC01

INTERVENTIONS:
Biological: anticancer medication A01; immune cells IC01 — The administration of the anticancer medication A01 and immune cells IC01 will be performed in The Second Hospital of Jiaxing, Zhejiang, China.
  The subjects will be observed for any side effects during this time and all the adverse events will be recorded.

SUMMARY:
This is an open-label study to evaluate the safety and efficacy of an anticancer medication (A01) combined with immune cells (IC01) in subjects with advanced Gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to any research procedures;
2. Age: 18 Years to 70 Years;
3. The patient's biological parent or child whose age ≥18 years voluntarily donates peripheral blood (200 ml) for the treatment, and who signs the informed consent form independently;
4. Histologically confirmed diagnosis of gastrointestinal cancer;
5. Patients who have received at least one standard treatment (surgery, chemotherapy, radiotherapy, or targeted therapy) or refuse to receive standard treatments;
6. Karnofsky Performance Status (KPS) score ≥ 70
7. Expected survival ≥ 3 months
8. Adequate organ function defined as: ANC≥3.5×10^9/L, PLT≥50×10^9/L, ALB≥25g/L, AST≤2.5×ULN, ALT≤2.5×ULN, TBIL≤1.5×ULN
9. If a subject is a female of childbearing potential, she must have a negative urine pregnancy test result.

Exclusion Criteria:

1. Patients who received chemotherapy, large-field radiotherapy or participated in other studies of anti-tumor therapy within 2 weeks before enrollment;
2. Patients who have not recovered from adverse reactions related to above-mentioned procedures;
3. Patients with two types of primary solid tumors;
4. Patients with brain metastases or bone metastases;
5. Patients with poorly controlled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 90 mmHg), or cardiovascular and cerebrovascular diseases with clinical significance, such as cerebrovascular accident (within 6 months before signing informed consent), myocardial infarction (within 6 months before signing informed consent), unstable angina, congestive heart failure (New York Heart Association Class II or above), or severe arrhythmia which can't be controlled with drugs or have potential impact on treatment;
6. Patients with other serious organic diseases or mental disorders;
7. Patients with systemic or active infection;
8. Patients with positive HIV test result;
9. Patients who have received an organ transplant;
10. Patients who are breastfeeding or pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with infusion of the anticancer medication or the immune cells will be assessed. | Day 0 to 4 months after the end of the trial
  Incidence and duration of all the adverse events will be recorded. The severity of adverse events will be evaluated according to NCI-CTCAE v4.03 criteria.

SECONDARY OUTCOMES:
Tumor Response of the treatment in patients with advanced gastrointestinal cancer. | Before treatment and Day 28 to 4 months after the end of the treatment
  Response Evaluation Criteria in Solid Tumors (RECIST) from the NCI will be used for assessment of radiographic response.

IPD SHARING:
Plan to Share IPD: No